CLINICAL TRIAL: NCT04921384
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate Efficacy and Safety of Eptinezumab for the Preventive Treatment of Migraine
Brief Title: Eptinezumab as Preventive Treatment of Migraine in Adults With Migraine
Acronym: Sunrise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19140A; 2020-001657-42 (EudraCT Number)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eptinezumab 300 mg (Experimental): 300 mg eptinezumab by intravenous (IV) infusion.
  Interventions: Drug: Eptinezumab
- Eptinezumab 100 mg (Experimental): 100 mg eptinezumab by IV infusion.
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Placebo by IV infusion.
  Interventions: Drug: Placebo; Drug: Eptinezumab

INTERVENTIONS:
Drug: Placebo — 0.9% normal saline, intravenously
  Arms: Placebo
Drug: Eptinezumab — Solution for infusion, intravenously
  Other Names: Lu AG09221

SUMMARY:
This study evaluates the efficacy of eptinezumab to prevent migraine in participants with chronic migraine.

DETAILED DESCRIPTION:
This is an interventional, multi-regional, multi-site, randomized, double-blind, placebo-controlled Phase III study, to confirm the efficacy and safety of eptinezumab in participants with chronic migraine who are eligible for preventive treatment.

participants will be randomly allocated to one of three treatment groups: eptinezumab 300 mg, eptinezumab 100 mg, or placebo.

The double-blind, placebo-controlled treatment period will be followed by an extension period where all participants will receive active treatment to further assess the safety and tolerability of eptinezumab.

The total study duration from the Screening Visit to the Safety Follow-up Visit is approximately 36 weeks and includes a Screening Period (28-30 days), a Placebo-controlled Period (12 weeks), an Extension Period (12 weeks), and a Safety Follow-up Period (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of CM as defined by IHS ICHD-3 guidelines confirmed at screening visit with a history of migraine onset at least 12 months prior to the Screening Visit.
* The participant has a migraine onset at ≤50 years of age.
* The participant has ≥8 migraine days per month for each month within the past 3 months prior to the Screening Visit.
* The participant fulfils the following criteria for migraine in prospectively collected information in the eDiary during the screening period:
* Migraine occurring on ≥8 days and headache occurring on ≥15 to ≤26 days.
* The participant has demonstrated compliance with the Headache eDiary by entry of data for at least 24 of the 28 days following the Screening Visit.
* The participant is aged ≥18 (≥20 for Taiwan) and ≤75 years at the Screening Visit.

Exclusion Criteria:

* The participant has received any medication targeting the calcitonin gene-related peptide (CGRP) pathway as preventive treatment of migraine.
* The participant has confounding and clinically significant pain syndromes, (for example, fibromyalgia, chronic low back pain, complex regional pain syndrome).
* The participant has a diagnosis of acute or active temporomandibular disorder.
* The participant has a history or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), ophthalmoplegic migraine, migraine with brainstem aura and migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration).
* The participant has a lifetime history of psychosis, bipolar mania, or dementia.
* Participants with other psychiatric conditions whose symptoms are not controlled or who have not been adequately treated for a minimum of 6 months prior to screening are also excluded.
* The participant has a history of clinically significant cardiovascular disease, including uncontrolled hypertension, vascular ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of monthly migraine days (MMDs) (Weeks 1-12) | Weeks 1-12

SECONDARY OUTCOMES:
Response: ≥50% reduction from baseline in MMDs (Weeks 1-12) | Weeks 1-12
Response: ≥75% reduction from baseline in MMDs (Weeks 1-4) | Weeks 1-4
Response: ≥75% reduction from baseline in MMDs, (Weeks 1-12) | Weeks 1-12
Migraine rate on the day after dosing | Day 1
Response: ≥50% reduction from baseline in monthly headache days (MHDs) (Weeks 1-12) | Weeks 1-12
Change from baseline in the number of MHDs (Weeks 1-12) | Weeks 1-12
Response: ≥75% reduction from baseline in MHDs (Weeks 1-4) | Weeks 1-4
Change from baseline in rate of migraines with severe pain intensity (Weeks 1-12) | Weeks 1-12
Change from baseline in rate of headaches with severe pain intensity (Weeks 1-12) | Weeks 1-12
Change from baseline in the number of MMDs with use of acute medication (Weeks 1-12) | Weeks 1-12
Patient Global Impression of Change (PGIC) score at week 12 | Week 12
Most Bothersome Symptom (MBS) score at Week 12, as measured relative to Screening | Screening to Week 12
Change from baseline to Week 12 in the Headache Impact Test (HIT-6) score | Baseline to Week 12
Change from baseline to Week 12 in the Migraine-Specific Quality of Life (MSQ v2.1) sub-scores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) | Baseline to Week 12
Change from baseline to Week 12 in the Health-Related Quality of Life (EQ-5D-5L) Visual Analogue Scale (VAS) score | Baseline to Week 12
Health Care Resources Utilization (HCRU) | Baseline to Week 12
  Migraine-specific healthcare resource utilization information will be collected in terms of outpatient health care professional visits, emergency room visits, hospital admissions, as well as duration of hospital stays.
Change from baseline to Week 12 in the Work Productivity and Activity Impairment Questionnaire: Migraine (WPAI:M) sub-scores (Absenteeism, Presenteeism, Work productivity loss, Activity impairment) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (87):
- China (15):
  - The First Medical Center of The Chinese PLA General Hospital (301 Hospital), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University - Yanjiang Campus, Guangzhou, Guangdong
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University - Main Campus, Wuhan, Hubei
  - Beijing Chaoyang Hospital Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Affiliated Hospital With Nanjing Medical University(Jiangsu Province Hospital), Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Norman Bethune Hospital of Jilin University - Ziqiang Campus, Changchun
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Georgia (7):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center -3 Nakalakevis Kucha, Tbilisi
  - Ltd Israel-Georgia Medical Research Clinic Helsicore, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - Aversi Clinic LTD, Tbilisi
  - MediClubGeorgia Ltd, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
  - S. Khechinashvili University Clinic, Ltd., Tbilisi
- Japan (27):
  - Tokyo Dental College Ichikawa General Hospital, Ichikawa-Shi, Chiba
  - Nakamura Memorial Hospital, Sapporo-Shi Chuo-Ku, Hokkaidô
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Sendai Headache and Cranial Nerves Clinic, Sendai-Shi Taihaku-Ku, Miyagi
  - Makabe Clinic, Okayama-Shi Kita-Ku, Okayama-ken
  - Saitama Neuropsychiatric Institute, Saitama-shi, Saitama
  - Moriyama Neurological Center Hospital, Edogawa-ku, Tokyo
  - Shinagawa strings clinic, Minato-Ku, Tokyo
  - USUDA CLINIC for internal medicine, Setagaya-ku, Tokyo
  - Fukuuchi Pain Clinic, Shinjuku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Suzuki Kei Yasuragi clinic, Tachikawa-Shi, Tokyo
  - Nagamitsu Clinic, Hōfu, Yamaguchi
  - DOI Clinic Internal Medicine, Hirosima Naka-ku
  - Atsuchi Neurosurgery Hospital, Kagoshima
  - Ikeda Neurosurgical Clinic, Kasuga
  - Jinnouchi Neurosurgery Clinic, Kasuga-shi
  - Shin Matsudakai Atago Hospital, Kochi
  - Tatsuoka Neurology Clinic, Kyoto Shimojo-ku
  - Dokkyo Medical University Hospital, Mibu-Machi
  - Mito Kyodo General Hospital, Mito
  - Tominaga Hospital, Naniwa-ku
  - Tokyo headache clinic, Shibuya-ku
  - Japanese Red Cross Shizuoka Hospital, Shizuoka
  - Eiju General Hospital, Taitō City
  - Kitasato University Kitasato Institute Hospital, Tokyo
  - Toyota Memorial Hospital, Toyota-shi
- Poland (11):
  - Solumed Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim, Lesser Poland Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - ETG Zamosc - PPDS, Zamość, Lublin Voivodeship
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - ETG Neuroscience - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Gdynia - PRATIA - PPDS, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Silmedic Sp z o o, Katowice, Silesian Voivodeship
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice
  - Centrum Medyczne Kiepury Clinic, Sosnowiec
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Slovakia (4):
  - MUDr. Beata Dupejova, Neurologicka ambulancia, s.r.o., Banská Bystrica
  - IN MEDIC, s.r.o., Bardejov
  - KONZILIUM s.r.o, Dubnica nad Váhom
  - SANERA, s.r.o., Prešov
- South Korea (9):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggido
  - Chungnam National University Hospital, Daejeon
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

REFERENCES:
- [Derived] Yu S, Matsumori Y, Kim BK, Gryglas-Dworak A, Giorgadze G, Pozo-Rosich P, Krog Josiassen M, Ranc K, Ettrup A, Mittoux A, Sperling B, Takeshima T. Efficacy and safety of eptinezumab in a predominantly Asian population with chronic migraine: Results of the randomized, double-blind, placebo-controlled SUNRISE trial. Cephalalgia. 2025 Oct;45(10):3331024251386095. doi: 10.1177/03331024251386095. Epub 2025 Oct 15. PMID 41091746